CLINICAL TRIAL: NCT00015223
Title: Methyphendidate in the Treatment of Cocaine Dependent Patients With Adult ADHD
Brief Title: Methylphenidate in the Treatment of Cocaine Dependent Patients With Adult Attention Deficit Hyperactivity Disorder - 5
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: Cincinnati MDRU (Other)
Masking: Double | Purpose: Treatment
Other Study IDs: NIDA-5-0013-5; Y01-5-0013-5
Record Dates: First submitted 2001-04-18; First posted 2001-04-18 (Estimated); Last update posted 2017-01-16 (Estimated); Status verified 2012-10

CONDITIONS: Cocaine-Related Disorders; Substance-Related Disorders
MeSH Terms: conditions — Cocaine-Related Disorders; Substance-Related Disorders | interventions — Methylphenidate

INTERVENTIONS:
Drug: Methylphenidate

SUMMARY:
The purpose of this study is the use of Methylphenidate in the treatment of cocaine dependence and Attention Deficit Hyperactivity Disorder (ADHD) comorbidity.

DETAILED DESCRIPTION:
The objective of this study is to determine the safety and efficacy of methylphenidate in a population of patients who are cocaine dependent and suffer from attention deficit hyperactivity disorder.

ELIGIBILITY:
Inclusion Criteria:

Cocaine-dependent. Meets the DSM-IV criteria for ADHD. Actively using cocaine within the past 30 days of screening.

Exclusion Criteria:

Symptoms of AIDS. Significant medical disorder. DSM-IV criteria for any substance other than cocaine, alcohol, nicotine, marijuana, caffeine. Requires detoxification from ETOH or benzos. History of seizures.

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0
Dates: Start 1997-06; Primary Completion 1999-07 (Actual); Study Completion 1999-08 (Actual)

PRIMARY OUTCOMES:
Cocaine use
Methylphenidate retention
Safety assessments
Psychosocial counseling sessions

CONTACTS AND LOCATIONS:
Overall Officials: Gene Somoza, M.D., Principal Investigator — U of Cincinnati
Locations (1):
- Cincinnati MDRU, Cincinnati, Ohio, United States